CLINICAL TRIAL: NCT04120415
Title: EHVA T02 (European HIV Vaccine Alliance Therapeutic Trial 02)/ANRS VRI07: A Phase II Randomised, Placebo-controlled Trial of Vedolizumab With or Without Therapeutic HIV MVA Vaccine in Individuals Who Started Antiretrovirals During Primary or Chronic Infection
Brief Title: A HIV Vaccine Trial in Individuals Who Started Antiretrovirals During Primary or Chronic Infection (EHVA T02)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: EuroVacc Foundation (Other); European AIDS Treatment Group (EATG) (Unknown); Medical Research Council (Other Government); University College London Hospitals (Other); University of Liverpool (Other); Erasmus Medical Center (Other); Henri Mondor University Hospital (Other); European Georges Pompidou Hospital (Other); Saint-Louis Hospital, Paris, France (Other); Centre Hospitalier Universitaire Vaudois (Other); Chelsea and Westminster Hospital, UK (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other); Hospital Clinic of Barcelona (Other); Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS (Network); Imperial College London (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); European Commission (Other); Swiss Government (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EHVA T02/ANRS VRI07
Record Dates: First submitted 2019-09-30; First posted 2019-10-09 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Vaccines; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccine and Vedolizumab infusion (Experimental): Vaccine:
  The vaccine is MVA HIV-B which is a solution of HIV MVA vectors in S08 buffer (10mM Tris/hydrochloride (Tris/HCl), Saccharose 5% (w/v), 10mM Sodium Glutamate (Na Glu), 50mM Sodium Chloride (NaCl), water PPI, pH 8.0).
  Vedolizumab infusion (Entyvio):
  Vedolizumab (300mg) is administered as an intravenous infusion (255 ml).
  Interventions: Biological: Vaccine and vedolizumab (Entyvio)
- Placebo vaccine and Vedolizumab infusion (Experimental): Placebo vaccine:
  The placebo for MVA HIV-B to be used in this trial is a solution composed of S08 buffer (as for the MVA vaccine).
  Vedolizumab infusion (Entyvio):
  Vedolizumab (300mg) is administered as an intravenous infusion (255 ml)
  Interventions: Biological: Placebo vaccine and vedolizumab infusion (Entyvio)
- Placebo vaccine and placebo infusion (Placebo Comparator): Placebo vaccine:
  The placebo for MVA HIV-B to be used in this trial is a solution composed of S08 buffer (as for the MVA vaccine).
  Placebo infusion:
  Sodium Chloride (NaCl) 0.9% administered as an intravenous infusion (255ml)
  Interventions: Biological: Placebo vaccine and placebo infusion

INTERVENTIONS:
Biological: Vaccine and vedolizumab (Entyvio) — Vaccine and vedolizumab infusion (Entyvio):
  0.5ml of MVA HIV-B (1 x 108 pfu/ml) will be administered intramuscularly in the deltoid muscle of the non-dominant upper arm at weeks 0 and 8. Participants will be observed after the injection.
  Vedolizumab (300mg) is administered as an intravenous infusion (255 ml) over 30 mins in the dominant arm at weeks 10,12,16,20,24,28 and 32. After infusion, the line should be flushed with 30ml of normal saline. Participants will be observed throughout and after the infusion.
  Arms: Vaccine and Vedolizumab infusion
Biological: Placebo vaccine and vedolizumab infusion (Entyvio) — Placebo Vaccine:
  The placebo for MVA HIV-B to be used is a solution composed of S08 buffer (as for the MVA vaccine) that will be intramuscularly in the deltoid muscle of the non-dominant upper arm at weeks 0 and 8. Participants will be observed after the injection.
  Vedolizumab infusion (Entyvio):
  Vedolizumab (300mg) is administered as an intravenous infusion (255 ml) over 30 mins in the dominant arm at weeks 10,12,16,20,24,28 and 32. After infusion, the line should be flushed with 30ml of normal saline. Participants will be observed throughout and after the infusion.
  Arms: Placebo vaccine and Vedolizumab infusion
Biological: Placebo vaccine and placebo infusion — Placebo Vaccine:
  The placebo for MVA HIV-B to be used is a solution composed of S08 buffer (as for the MVA vaccine) that will be intramuscularly in the deltoid muscle of the non-dominant upper arm at weeks 0 and 8. Participants will be observed after the injection.
  Placebo infusion (Entyvio):
  255ml Sodium Chloride (NaCl) 0.9% bag administered as an intravenous infusion over 30 mins in the dominant arm at weeks 10,12,16,20,24,28 and 32. Participants will be observed throughout and after the infusion.
  Arms: Placebo vaccine and placebo infusion

SUMMARY:
EHVA T02 is an international, phase II, double-blind study to evaluate two experimental arms each compared to placebo control in HIV-1 positive participants to see if either has a clinically relevant impact on viral replication.

DETAILED DESCRIPTION:
Screening will take place during the 6 weeks prior to randomisation. Eligible participants will be enrolled at week 0 and randomised to MVA HIV-B vaccine followed by vedolizumab, vedolizumab + placebo vaccine, or placebo vaccine + placebo infusions.

Participants will be randomised at each centre through web-based randomisation after entering the eligibility criteria. There will be two strata: one for those who started treatment during primary infection, and one for those who started treatment during chronic infection.

69 eligible individuals from collaborating European Countries will be enrolled, aiming for approximately half who started cART in primary infection and half who started in chronic infection. Participants continue from the screening visit (up to 6 weeks before enrolment) to the last visit, a maximum of 60 weeks (around 14 months), although follow-up will continue through to the time when virus is fully suppressed.

Treatment will be interrupted at week 18 and resumed when the viral load is confirmed to have rebounded to ≥100,000 copies/ml, or the CD4 falls to ≤350 cells/mm3, confirmed, or there is evidence of disease progression, or they have completed 24 weeks of treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1-infected
2. Aged 18 - 65 years old on the day of screening
3. Weight >50kg
4. Willing and able to provide written informed consent
5. Nadir CD4 count > 300 cells/mm3
6. CD4 count at screening > 500 cells/mm3
7. Viral load <50 copies/ml at screening.
8. Started cART after 2009 and on cART for at least one year prior to screening
9. Willing to interrupt cART for up to 24 weeks and change cART regimen if required
10. If sexually active, willing to use a reliable method of reducing the risk of transmission to their sexual partners during treatment interruption (which could include PrEP for their sexual partners)
11. If heterosexually active and able to have children, willing to use a highly effective method of contraception with partner (combined oral contraceptive pill; injectable or implanted contraceptive; IUD/IUS; physiological or anatomical sterility (in self or partner) from 2 weeks before enrolment until 18 weeks after the last injection/infusion
12. If women of childbearing potential*, willing to undergo urine pregnancy tests prior to administration of an injection and an infusion
13. Willing to avoid all other vaccines within 4 weeks of scheduled study injections
14. Willing and able to comply with visit schedule and provide blood samples
15. Being covered by medical insurance or in National Healthcare System

    * A woman will be considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Exclusion Criteria:

1. Pregnant or lactating
2. HIV-2 infection (either isolated or associated with HIV-1)
3. VL >200 copies/ml on 2 occasions in the 12 months prior to screening
4. Previous interruptions in cART
5. Previous virological failures defined by loss of virological suppression with the presence of resistant mutations
6. Haemoglobin (Hb <12g/dL for males, <11g/dL for females)
7. Concomitant or previous conditions that preclude injection of vaccines/infusion of monoclonal antibody and PML in the past
8. History of experimental vaccinations against HIV
9. Previous treatment with chemotherapy (except for chemotherapy injected into skin lesions for Kaposi's sarcoma)
10. Treatment with systemic corticoids or immuno-suppressive agents ongoing or in the 12 weeks prior to randomisation in the trial
11. Received natalizumab or rituximab ever in the past
12. Received a TNF blocker in the past 60 days
13. Administration of an inactivated vaccine within 30 days or a live vaccine within 60 days prior to randomisation
14. Presence of a skin condition or marking that precludes inspection of the injection/infusion site
15. History of cancer (except basal cellular skin carcinoma or Kaposi's sarcoma)
16. History of significant neurological disease or cardiovascular disease (angina, myocardial infarction, transient ischemic attack, stroke); participants with controlled blood pressure are eligible
17. History of clinical autoimmune disease
18. Ongoing diseases including uncontrolled active severe infection, cardiac, pulmonary (excluding mild asthma), thyroid, renal or neurological (peripheral or central) diseases
19. Active or latent tuberculosis (unless prophylaxis in past as per local practice) - (participant must be screened for tuberculosis before starting infusions, according to routine practice)
20. Presence of pathogenic bacteria or parasites in faeces at screening
21. Participating in another biomedical research study within 30 days of randomisation
22. Known hypersensitivity to any component of the vaccine formulation used in this trial including eggs or have severe or multiple allergies to drugs or pharmaceutical agents, or any hypersensitivity to the active substance or to any of the excipients of vedolizumab.
23. Liver disease including hepatitis B (surface antigen positive) or hepatitis C (antigen or PCR positive)
24. A clinically significant abnormality on ECG
25. Hypernatraemia or hyperchloraemia
26. History of severe local or general reaction to vaccination defined as

    1. local: extensive, indurated redness and swelling involving most of the arm, not resolving within 72 hours
    2. general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
27. Grade 2 or worse routine laboratory parameters. Hyperbilirubinaemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Area under the HIV RNA curve | Time from treatment interruption (scheduled for 18 weeks after entering the trial) to 24 weeks post-treatment interruption
  Area under the HIV RNA curve from treatment interruption (scheduled for 18 weeks after entering the trial)

SECONDARY OUTCOMES:
Virological outcome measures | For participants commencing treatment interruption only, critical time points weeks 19 through to to week 42.
  Time from treatment interruption (scheduled for 18 weeks after entering the trial) to the earliest of reaching HIV RNA ≥ 100 000 copies/ml (confirmed on a separate sample) or resuming antiretroviral therapy for any reason over a period of 24 weeks.
Virological outcome measures | From randomisation to study completion about 54 weeks
  Level of HIV total RNA
Virological outcome measures | From randomisation to study completion about 54 weeks
  Cell Associated (CA) HIV RNA Quantification
Virological outcome measures | Time from treatment interruption, only in participants commencing treatment interruption, up to 24 weeks after ATI
  First local maximum (peak) level of HIV total RNA during treatment interruption
Virological outcome measures | Time from treatment interruption, only in participants commencing treatment interruption, up to 24 weeks after ATI
  Rate of increase of HIV total RNA between the last measure below the lower detection and the first local maximum
Virological outcome measures | Time from treatment interruption, only in participants commencing treatment interruption, up to 24 weeks after ATI
  Setpoint (two stable measures following a transient increase of HIV RNA)

OTHER OUTCOMES:
Safety outcome measures: Grade 3 or worse solicited clinical and laboratory adverse events | From randomisation to study completion about 54 weeks
  Occurrence of grade 3 or worse solicited clinical and laboratory adverse events
Safety outcome measures: Any adverse event leading to interruption in the vaccine/placebo or vedolizumab/placebo | From randomisation to study completion about 54 weeks
  Occurrence of any adverse event leading to interruption in the vaccine/placebo or vedolizumab/placebo
Safety outcome measures: Any event that results in resuming treatment during the ATI | Time form treatment interruption to resuming treatment, up to 24 weeks after ATI
  Occurrence of any event that results in resuming treatment during the ATI
Safety outcome measures: Serious Adverse Events | From randomisation until 30 days after the last protocol visit
  Occurrence of Serious Adverse Events
Safety outcome measures: Other clinical and laboratory adverse events | From randomisation to study completion about 54 weeks
  Occurrence of other clinical and laboratory adverse events
Safety outcome measures: Change in absolute CD4 | From randomisation to study completion about 54 weeks
  Observation of change in absolute CD4 count
Safety outcome measures: Time to VL suppression after restarting cART | From randomisation to VL suppression (= VL is undetectable (<50copies/ml)) after restarting cART until the participant returns to an undetectable viral load, about 54 weeks]
  Time to VL suppression after restarting cART
Exploratory Immunological outcome measures: Characterization of vaccine induced CD4 and CD8 T-cell produced cytokine profile | From randomisation to study completion about 54 weeks
  Observation of vaccine induced CD4 and CD8 T-cell produced cytokines by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Yves Levy, MD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (4):
- France (2):
  - Service Immunologie clinique et maladies infectieuses, Hôpital Henri Mondor, Paris, Creteil
  - Hotel Dieu, Paris
- Centre d'Immunothérapie et Vaccinologie, CHUV, Lausanne, Canton of Vaud, Switzerland
- St Stephens Centre, Chelsea & Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No